CLINICAL TRIAL: NCT01380613
Title: The Impact of Neighborhoods, Networks, and Depression on Drug Users' HIV Risk
Brief Title: Neighborhoods, Networks, Depression, and HIV Risk
Acronym: Workshop
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Carl Latkin, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DESPR-DA022961-03; R01DA022961 (NIH)
Record Dates: First submitted 2011-03-07; First posted 2011-06-27 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: HIV; Depression; Drug Use
Keywords: HIV; depression; drug use,; risk reduction
MeSH Terms: conditions — Depression; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Workshop Control (Active Comparator): Participants receive HIV/STDs risk reduction information.
  Interventions: Behavioral: Workshop control
- Intervention Workshop (Experimental): Participants learn skills to cope with depressive symptoms and stress as well as safer sex and injection skills.
  Interventions: Behavioral: Workshop

INTERVENTIONS:
Behavioral: Workshop — 10 session intervention
  Arms: Intervention Workshop
Behavioral: Workshop control — 1 session intervention on standard HIV/STD information
  Arms: Workshop Control

SUMMARY:
The goal of this study is to examine how social networks, neighborhood, and depression are related to HIV risk. The intervention is designed to train individuals to cope with feelings of depression or stress as a way to reduce their risk for HIV.

DETAILED DESCRIPTION:
This study included implementation and evaluation of a small group, randomized controlled, phase II intervention to reduce depressive symptoms and HIV risk behaviors among inner city drug users. The intervention included elements of cognitive behavioral therapy (CBT) for depression among impoverished individuals, emphasizing depressive cognitions and behaviors theorized to be associated with depression and with HIV risk behaviors among mildly to moderately depressed drug users. In addition, the study examined active drug users' social and environmental pathways to depression and subsequent HIV risk behaviors. Specifically, we will hypothesized mediating/moderating effects of neighborhood characteristics, social network factors, and individual level factors on depressive symptoms and HIV risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. 18-55 years old
2. HIV Risk Behavior:

3a. Injected drugs more than 3 times in the past week OR

3b. Snorted/sniffed heroin or cocaine or smoked crack in the past 6 months AND had 1 of the following sex risks in the past 6 months: i) 2 or more sex partners ii) Had a sex partner who injected drugs iii)Had a sex partner who smoked crack iv) Had a sex partner who was HIV+

4. Willingness to attend group sessions

Exclusion Criteria:

1. Enrolled in another HIV behavioral intervention or depression study in past the 3 years
2. Enrolled in another Lighthouse study in past the 5 years
3. Enrolled in the formative research (Phase 1) or pilot (Phase 2) of the current project.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 965 (Actual)
Dates: Start 2007-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Depressive Symptoms Measured by the CESD Scale at 6 months | 6 months
Change from Baseline in Depressive Symptoms Measured by the CESD Scale at 12 months | 12 months

SECONDARY OUTCOMES:
Change from Baseline in Sex Risk Behavior Based on Number of Sex Partners and Condom Use at 6 months | 6 months
Change from Baseline in Injection Risk Behavior Based on Sharing Needles, Cookers, and Cotton For Injection and Drug Splitting at 6 months | 6 months
Change from Baseline in Sex Risk Behavior Based on Number of Sex Partners and Condom Use at 12 months | 12 months
Change from Baseline in Injection Risk Behavior Based on Sharing Needles, Cookers, and Cotton For Injection and Drug Splitting at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Latkin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Lighthouse Studies @ Peer Points- JHSPH, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Tobin K, Davey-Rothwell MA, Nonyane BAS, Knowlton A, Wissow L, Latkin CA. RCT of an integrated CBT-HIV intervention on depressive symptoms and HIV risk. PLoS One. 2017 Dec 14;12(12):e0187180. doi: 10.1371/journal.pone.0187180. eCollection 2017. PMID 29240757